CLINICAL TRIAL: NCT02044575
Title: Clock Genes in Patients With Refractory Septic Shock (SeptiClock) - Pilot Study
Status: Completed | Type: Observational
Sponsor: Claudia Spies (Other)
Responsible Party: Sponsor-Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine, CVK/CCM, Charité - University Medicine Berlin, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: SeptiClock
Record Dates: First submitted 2014-01-20; First posted 2014-01-24 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Septic Shock
Keywords: Clock genes, circadian regulation
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Critically ill patients: Intensive care unit patients with refractory septic shock

SUMMARY:
Despite large efforts trying to improve diagnostic and therapy of sepsis have been made over the last decade (e.g. initiation of the Surviving Sepsis Campaign, defining evidence based sepsis therapy bundles) the mortality of septic shock remains high and causes high socioeconomical burden of disease.

The purpose of this pilot study is to evaluate the design and conduct of a projected full scale clinical trial.

DETAILED DESCRIPTION:
A functional clock is required for induction of several proinflammatory genes, not shown in septic patient settings, yet.

Clock genes are involved in modulating the activity of several transcription factors that are important regulators of immune functions (e.g. HIF1-α, STAT1, STAT3, and NF-κB) (Bellet MM et al., 2013).

Furthermore, polymorphisms such as rs7221412, a common polymorphism near period homolog 1 (PER1), was associated with the timing of activity rhythms and also showed a suggestive time-dependent relationship with both cerebral cortex and monocytes PER1 expression and an association with time of death (Lim ASP et al., 2012).

This explorative project is a pilot study. First data are generated for the assessment of the circadian system in patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with age 18 years and above,
* Patient at intensive care units (8i, 9i and 1i at Charité - University Medicine Berlin , Campus Virchow- Klinikum),
* Septic shock (ACCP/SCCM (American College of Chest Physicians/Society of Critical Care Medicine) consensus definitions) AND Norepinephrine dosage of >0.3 μg/kg/min for at least 2 hours

Exclusion Criteria:

* Pregnant or lactating female patient,
* Participation in another interventional study (30 days before study inclusion and during study participation),
* Acute leucemia,
* Severe leukocytosis (>50,000/nl),
* Severe thrombocytopenia (<5,000/nl),
* Autoimmune disease with systemic medication of ≥10 mg prednisolone equivalent or previous transplantation,
* Patients receiving interferon therapy (last 14 days),
* Patients with known hypersensitivity GM-CSF or known antibodies against GM-CSF, yeast-derived products or any component of the study medication,
* Ongoing (concomitant) chemotherapy or radiotherapy for malignancy,
* Acute pulmonary embolism or acute myocardial infarction within last 72 hours,
* Cardiopulmonary resuscitation within last 7 days,
* Moribund patient (life expectancy <72 hrs.),
* Presence of a do-not-resuscitate or do-not-intubate order,
* Known human immunodeficiency virus (HIV) infection or chronic viral hepatitis
* Lacking willingness to save and hand out data within the study
* Accommodation in an institution due to an official or judicial order
* The informed consent of the patient or the subject's legally acceptable representative can´t be obtained in time
* Patient has a power of attorney or patient's provision, where he/she refuses participation in any clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with septic shock
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-01-21 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Assessment of circadian regulation | These parameters are measured during intensive care unit stay, for a maximum of 3 days
  Circadian regulation by expression of clock genes

SECONDARY OUTCOMES:
Time on mechanical ventilation | They are followed up until the end of intensive care unit stay - or, for a maximum of 28 days
Intensive care unit length of stay | Participants will be followed for the duration of intensive care stay, an expected average of 4 weeks
Hospital length of stay | Participants will be followed for the duration of intensive care stay, an expected average of 5 weeks
Simplified Acute Physiology Score (SOFA II) | They are measured until the end of intensive care unit stay - or, for a maximum of 28 days.
Sequential Organ Failure Assessment (SOFA) | They are measured until the end of intensive care unit stay - or, for a maximum of 28 days.
Therapeutic Intervention Scoring System (TISS-28) | They are measured until the end of intensive care unit stay - or, for a maximum of 28 days.
Mortality | 6 months after intensive care unit discharge
Light frequencies | Light frequencies are measured until the end of intensive care unit stay - or, for a maximum of 28 days
Light levels (lux) | Light levels are measured until the end of intensive care unit stay - or, for a maximum of 28 days
Cortisol | This parameter is measured in ng/ml during intensive care unit stay, for a maximum of 3 days
Melatonin | This parameter is measured in pg/ml during intensive care unit stay, for a maximum of 3 days
Quality of life | Up to 3 and 6 months
  Quality of life is measured by SF-36 questionnaire
Cognitive function | Up to 3 and 6 months
  Cognitive function is measured by Repeatable Battery for the Assessment of Neuropsychological Status
Multiplex-Genexpression analysis | These parameters are measured during intensive care unit stay, for a maximum of 3 days
  Ncounter neuroinflammation and micro rna panel are analysed

OTHER OUTCOMES:
Nagalase enzyme activity | This parameter is measured at the beginning of the investigation
  Nagalase Enzyme activity is expressed in nmol/min per Milliliter. Analysis is evaluated with the perioperative Nagalase results of 10 patients in the clinical trial Phydelio (EudraCT-No 2008-007237-47).
Venous return | This parameter is measured at the beginning of the investigation
  Venous return will be assessed after ICU admission by venous return pressure gradient (dVR)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Campus Charité Mitte and Campus Virchow - Klinikum, Charité- Universitätsmedizin, Berlin, Germany

REFERENCES:
- [Background] Bellet MM, Deriu E, Liu JZ, Grimaldi B, Blaschitz C, Zeller M, Edwards RA, Sahar S, Dandekar S, Baldi P, George MD, Raffatellu M, Sassone-Corsi P. Circadian clock regulates the host response to Salmonella. Proc Natl Acad Sci U S A. 2013 Jun 11;110(24):9897-902. doi: 10.1073/pnas.1120636110. Epub 2013 May 28. PMID 23716692
- [Background] Lim AS, Chang AM, Shulman JM, Raj T, Chibnik LB, Cain SW, Rothamel K, Benoist C, Myers AJ, Czeisler CA, Buchman AS, Bennett DA, Duffy JF, Saper CB, De Jager PL. A common polymorphism near PER1 and the timing of human behavioral rhythms. Ann Neurol. 2012 Sep;72(3):324-34. doi: 10.1002/ana.23636. PMID 23034908
- [Derived] Lachmann G, Ananthasubramaniam B, Wunsch VA, Scherfig LM, von Haefen C, Knaak C, Edel A, Ehlen L, Koller B, Goldmann A, Herzel H, Kramer A, Spies C. Circadian rhythms in septic shock patients. Ann Intensive Care. 2021 Apr 26;11(1):64. doi: 10.1186/s13613-021-00833-5. PMID 33900485